CLINICAL TRIAL: NCT06353022
Title: Minimal Residual Disease-based Strategy with T-Cell Redirector After Treatment with Daratumumab, Bortezomib, Lenalidomide, and Dexamethasone (D-VRd) in Newly Diagnosed Multiple Myeloma: a Phase 2 (IFM 2022-01)
Brief Title: Minimal Residual Disease-based Strategy with T-Cell Redirector After Treatment with Daratumumab, Bortezomib, Lenalidomide, and Dexamethasone (D-VRd) in Newly Diagnosed Multiple Myeloma
Acronym: IFm2022-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC23_0267; 2023-508310-41 (EudraCT Number)
Record Dates: First submitted 2024-03-22; First posted 2024-04-08 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Newly Diagnosed; Teclistamab; Talquetamab
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab; Lenalidomide; Bortezomib; daratumumab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Teclistamab and Lenalidomide (Experimental): Patients treated with Teclistamab and Lenalidomide for finite duration.
  Interventions: Drug: Teclistamab; Drug: Lenalidomide; Drug: Bortezomib; Drug: Daratumumab; Drug: Dexamethasone
- Talquetamab andTeclistamab (Experimental): Patients treated with Teclistamab and Talquetamab for finite duration
  Interventions: Drug: Teclistamab; Drug: Talquetamab; Drug: Lenalidomide; Drug: Bortezomib; Drug: Daratumumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Teclistamab — Maintenance therapy wtih teclistamab (administered via SC injections) for finite duration. Teclistamab will be used in 28 day cycles following initial step up doses
  Other Names: No more information
Drug: Talquetamab — Maintenance therapy with talquetamab (administered via SC injections) for finite duration. Talquetamab will be used in 28 day cycles following initial step up doses
  Other Names: No more information
  Arms: Talquetamab andTeclistamab
Drug: Lenalidomide — Induction therapy with lenalidomide:
  Lenalidomide 25 mg/day oral from Day 1 to Day 21.
  Maintenance therapy lenalidomide (administered orally) for finite duration.
  Other Names: No more information
Drug: Bortezomib — Induction therapy with Borthezomib Cycle 1 to 6: Bortezomib 1.3 mg/m² SC twice a week on Days 1, 4, 8 and 11
  Other Names: No more information
Drug: Daratumumab — Induction therapy with Daratumumab Cycle 1 to 6 Daratumumab 1800 mg SC on Days 1, 8, 15, 22 of Cycle 1 and Cycle 2 and on Days 1 and 15 of Cycle 3
  Other Names: No more information
Drug: Dexamethasone — Induction therapy with Dexamethasone:
  cycle 1 to 3 Dexamethasone 40 mg/day oral or IV on Days 1, 8, 15, 22 Cycle 4 to 6 --> Dexamethasone 40 mg/day oral or IV on Days 1, 8, 15, 22
  Other Names: No more information

SUMMARY:
This is a Phase 2 study, open-label, 2-cohort, multicenter, national, interventional in patients with newly diagnosed multiple myeloma. The study will investigate teclistamab (Tec) in combination with lenalidomide (Len) (Tec-Len; Cohort A) or in combination with talquetamab (Tal) (Tec-Tal; Cohort B), allocated based on minimal residual disease (MRD) status (MRD [-] [standard-risk] vs MRD [+] [high-risk] respectively).

The patient population will consist of adults men and women at least 18 years to younger than 66 years of age, who meet eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

Each potential patient must satisfy all of the following criteria to be enrolled in the study:

Age, Type of Patient, Disease Characteristics

1. Male or female patients must be at least 18 years of age at the time of consent younger than 66 years.
2. Documented multiple myeloma satisfying the calcium elevation, renal insufficiency, anemia, and bone lesions (CRAB) criteria and measurable disease (Source: Rajkumar 2014)
3. Newly diagnosed patients eligible for high dose therapy and autologous Stem cell therapy.
4. Have a Karnofsky performance status score ≥50% (Eastern Cooperative Oncology Group ECOG performance status ECOG score ≤2.
5. Have clinical laboratory values meeting the following criteria.

   Sex and Contraceptive/Barrier Requirements
6. A female patient of childbearing potential must have a negative serum pregnancy test within 10 to 14 days prior to the start of study treatment and again either a serum or urine pregnancy test within 24 hours of the start of study treatment and must agree to further serum or urine pregnancy tests during the study and for a period of 6 months after the last dose of study treatments.
7. A female patient must be :

   1. Not of childbearing potential, or
   2. Of childbearing potential and 1) Practicing 2 reliable methods of contraception simultaneously including one highly effective method of contraception and one other effective method of contraception starting 4 weeks prior to dosing, throughout the study including during dose interruptions and for period of 6 months after the last dose of study treatments. For patients who are of childbearing potential.
8. A female patient must agree not to donate eggs or freeze for future use, for the purposes of assisted reproduction during the study and for a period of 6 months after the last dose of other study treatments. Female patients should consider preservation of eggs prior to study treatment as anti-cancer treatments may impair fertility.
9. A male patient must wear a condom (with spermicidal foam/gel/film/cream/suppository) when engaging in any activity that allows for passage of ejaculate to another person during the study and for a period of 6 months after the last dose of study treatments. If the male patient's partner is a female of childbearing potential, she must also be practicing a highly effective method of contraception.
10. A male patient must agree not to donate sperm for the purpose of reproduction during the study and for a period of 6 months after receiving the last dose of study. Male patients should consider preservation of sperm prior to study treatment as anti cancer treatments may impair fertility.

    Informed Consent
11. Voluntary written informed consent must be given before performance of any study related procedure not part of normal medical care, with the understanding that the patient may withdraw consent at any time without prejudice to future medical care.
12. Willing and able to adhere to the lifestyle restrictions specified in this protocol.
13. Affiliation with French social security system or beneficiary from such system.

Non inclusion Criteria:

Medical Conditions

1. Peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by the NCI CTCAE Version 5.0.
2. Chronic Obstructive Pulmonary Disease (COPD) with a Forced Expiratory Volume 1 (FEV1) <50% of predicted normal. Note that FEV1 testing is required for patients with known or suspected of having COPD or asthma and patients must be excluded if FEV1 <50% of predicted normal.
3. Moderate or severe persistent asthma within the past 2 years, uncontrolled asthma of any classification. Note that FEV1 testing is required for patients known or suspected asthma and patients must be excluded if FEV1 <50% of predicted normal.
4. Central Nervous System (CNS) involvement or clinical signs of meningeal involvement of multiple myeloma. If either is suspected, negative whole brain MRI and lumbar cytology are required.
5. Plasma cell leukemia, Waldenström's macroglobulinemia, polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes (POEMS) syndrome (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes), or primary light chain amyloidosis.
6. Any ongoing myelodysplastic syndrome or B cell malignancy (other than multiple myeloma).
7. Any history of malignancy, other than multiple myeloma, which is considered at high risk of recurrence requiring systemic therapy.
8. Active malignancies other than multiple myeloma. The only allowed exceptions are malignancies treated within the last 24 months that are considered cured:

   1. Non-muscle invasive bladder cancer.
   2. Non-melanoma skin cancers treated with curative therapy or localized melanoma treated with curative surgical resection alone
   3. Noninvasive cervical cancer
   4. Localized prostate cancer with a Gleason Score ≤7a, treated locally only
   5. Breast cancer: adequately treated lobular carcinoma in situ or ductal carcinoma in situ, or history of localized breast cancer
   6. Other malignancy that is considered cured with minimal risk of recurrence in consultation with the Sponsor
9. Stroke, transient ischemic attack, or seizure within 6 months prior to signing informed consent form.
10. Presence of the following cardiac conditions:

    1. New York Heart Association stage III or IV congestive heart failure
    2. Myocardial infarction or coronary artery bypass graft ≤6 months prior to enrollment
    3. History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
    4. Uncontrolled cardiac arrhythmia or clinically significant ECG (Electrocardiogram) abnormalities
    5. History of severe non-ischemic cardiomyopathy
11. Concurrent medical or psychiatric condition or disease that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study, such as:

    1. Acute diffuse infiltrative pulmonary disease
    2. Evidence of active systemic viral, fungal, or bacterial infection, requiring systemic antimicrobial therapy
    3. History of autoimmune disease with the exception of vitiligo, type I diabetes, and prior autoimmune thyroiditis that is currently euthyroid based on clinical symptoms and laboratory testing.
    4. Disabling psychiatric conditions, severe dementia, or altered mental status.
    5. Any other issue that would impair the ability of the patient to receive or tolerate the planned treatment at the investigational site, to understand informed consent or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient or that could prevent, limit, or confound the protocol- specified assessments.
    6. History of noncompliance with recommended medical treatments
12. Contraindications or life-threatening allergies, hypersensitivity, or intolerance to any study drug (daratumumab, bortezomib, lenalidomide, dexamethasone, teclistamab or talquetamab) or its excipients or analogues and study-required co-medication.
13. Incidence of gastrointestinal disease that may significantly alter the absorption of oral drugs.

    Prior/Concomitant Therapy
14. Prior or current systemic therapy or SCT for any plasma cell dyscrasia, with the exception of emergency use of a short course of corticosteroids before treatment.
15. Received a strong CYP3A4 inducer within 5 half-lives prior to the first dose of study treatment (Flockhart 2016: http://medicine.iupui.edu/flockhart/).
16. Plasmapheresis within 28 days prior to the first dose of study treatment.
17. Patient had major surgery or had significant traumatic injury within 2 weeks prior to the start of administration of study treatment, or will not have fully recovered from surgery, or has major surgery planned during the time the patient is expected to be treated in the study or within 2 weeks after administration of the last dose of study treatment.
18. Taken any disallowed therapies, Concomitant Therapy before the planned first dose of study intervention.
19. Received a live, attenuated vaccine within 4 weeks before the first dose of study drug. Non-live or replicating vaccines authorized for emergency use (eg, COVID-19) are allowed.

    Diagnostic Assessments
20. HIV infection (positive, history, treatment for HIV).
21. Hepatitis B infection (ie, HBsAg or HBV-DNA positive). In the event the infection status is unclear, quantitative viral levels are necessary to determine the infection status.
22. Active hepatitis C infection as measured by positive HCV-RNA testing. Patients with a history of HCV antibody positivity must undergo HCV RNA testing. If a patient with history of chronic hepatitis C infection (defined as both HCV antibody and HCV RNA positive) completed antiviral therapy and has undetectable HCV-RNA 12 weeks following the completion of therapy, the patient is eligible for the study.

    Other non-inclusions
23. Patients unable to complete baseline next generation sequencing (NGS) evaluation at Screening.
24. Patient is pregnant, a nursing mother, or planning to become pregnant while enrolled in this study or within 6 months after the last dose of study treatment.
25. Patient plans to father a child while enrolled in this study or within 6 months after the last dose of study treatment, whichever is later.
26. Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient or that could prevent, limit, or confound the protocol-specified assessments.
27. Person under guardianship, trusteeship or deprived of freedom by a judicial or administrative decision.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 103 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-04-26 (Estimated); Study Completion 2030-06-26 (Estimated)

PRIMARY OUTCOMES:
Rate of sustained MRD negativity (NGS, 10^-5) | 38 months
Rate of conversion from positive MRD to negative MRD (NGS, 10^-5) | 38 months

SECONDARY OUTCOMES:
Number of adverse events | 50 months
Rate of sustained MRD negativity (NGS, 10^-6) | 38 months
Rate of conversion from positive MRD to negative MRD (NGS, 10^-6). | 38 months
Rate of conversion from positive MRD to negative MRD (NGS, 10^-5). | 23 months
Number of the death | 74 months
Number of responses | 50 months
Number of progression-free survival | 74 months
Percentage of duration of response | 74 months
Percenatge of time to response | 74 months

OTHER OUTCOMES:
Percentage of value of biological prognostic factors influencing outcome and response. | 38 months
Percentage of score of quality of life | 38 months

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CH de la Côte Basque, Bayonne
  - CHU Caen, Caen
  - CHRU DIjon, Dijon
  - Chd Vendee, La Roche-sur-Yon
  - CHRU LILLE - Hôpital Claude Huriez, Lille
  - CHU Limoges, Limoges
  - CH Lyon Sud, Lyon
  - IPC Marseille Institut Paoli Calmettes, Marseille
  - CHU Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - APHP Hôpital Saint Louis, Paris
  - APHP Hôpital Saint-Antoine, Paris
  - APHP Hôpital La Pitié Salpétrière, Paris
  - CHU BORDEAUX - Hôpital du Haut Lévêque, Pessac
  - CHU Poitiers, Poitiers
  - CHRU Rennes - Hôpital de Pontchaillou, Rennes
  - ICANS Institut de Cancérologie Strasbourg Europe, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours Hôpital Bretonneau, Tours
  - CHRU Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy